CLINICAL TRIAL: NCT01814488
Title: A Phase II Multicentre Open-label Study on Allogeneic Stem Cell Transplantation From Unrelated, Cord-blood and Family Haploidentical Donors in Patients With Active Acute Leukemia
Brief Title: A Phase II Study on Allogeneic Stem Cell Transplantation in Patients With Active Acute Leukemia
Acronym: Gandalf-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004008-37 Gandalf-01
Record Dates: First submitted 2013-03-14; First posted 2013-03-20 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Acute Leukemia
Keywords: Active acute leukemia; PIF; Allogeneic transplant; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Marrow Unrelated Donor; Cord Blood; Family Haploidentical donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogenic transplant (Experimental): The experimental treatment consists in the application of a therapeutic strategy of allogeneic transplantation as a potential curative procedure in a population of patients with chemoresistant acute leukemias. Therapeutic intervention, namely the conditioning regimen as well as GVHD prophylaxis, are based on regimens currently in standard use in the context of allogeneic transplantation.
  Interventions: Procedure: allogeneic transplant

INTERVENTIONS:
Procedure: allogeneic transplant — Allogenic transplant using either a Marrow Unrelated Donor or a Cord Blood unit or a family Haploidentical donor.
  The conditioning regimen in standard use is:
  Thiotepa (Tepadina) i.v. 5 mg/kg/daily (total dose 10 mg/kg) day -7 and -6;
  Busulfan (Busilvex) i.v. 3,2 mg/kg/day (total dose 9,6 mg/kg) as a single daily dose day -5, -4, -3;
  Fludarabine i.v. 50 mg/m2 (total dose150 mg/m2) day -5, -4, -3.
  Primary antifungal prophylaxis is Micafungin 50 mg/die i.v. (1 mg/kg if <40 kg) day 0 to engraftment. After engraftment continue antifungal prophylaxis according to local practice.
  Other Names: Marrow Unrelated or Cord Blood or family Haploidentical donor

SUMMARY:
The experimental treatment consists in the application of a therapeutic strategy of allogeneic transplantation as a potential curative procedure in a population of patients with chemoresistant acute leukemias.

Therapeutic intervention, namely the conditioning regimen as well as GVHD prophylaxis, are based on regimens currently in standard use in the context of allogeneic transplantation.

DETAILED DESCRIPTION:
The experimental treatment consists in the application of a therapeutic strategy of allogeneic transplantation using either a Marrow Unrelated Donor (MUD) or a Cord Blood (CB) unit or a family Haploidentical (Haplo) donor as a potential curative procedure in a population of patients with chemoresistant acute leukemias for increase the overall survival in this patients.

Therapeutic intervention, namely the conditioning regimen as well as GVHD prophylaxis, are based on regimens currently in standard use in the context of allogeneic transplantation.

The Data Safety Monitoring Board (DSMB) in collaboration with the Steering Committee (SC) will make periodic monitoring to ensure the safety of patients enrolled in to the study. In particular, DSMB will check the periodic safety reports of serious adverse events, the primary or secondary graft failure and treated related mortality (TRM) data generated by the Data Management Center. A safety report will be generated every 30 enrolled patients completed 100 days of follow-up.

The population for analysis in the trial will be the Intention to Treat (ITT) population. All patients enrolled in the study will be included in the ITT analysis.

This study will explore the feasibility, safety and efficacy of allogeneic stem cell transplantation from unrelated, cord-blood and haploidentical donor in patients with an active leukemia. Due to the lack of detailed information from literature and the absence of alternative curative options in this patient population, criteria for sample size assessment do not refer to a formal statistical power calculation. Therefore, GITMO will promote enrollment of all patients with active leukemia eligible to allogeneic SCT in all Italian centres with the aim to collect outcome variables in ITT in the widest and most representative cohort of this specific patient population.

The choice of 80 patients transplanted is based on feasibility reasons and the expected patient population with these characteristics referred to the main Italian Transplant Centres in two year. GITMO survey data on transplant activity points to an estimated accrual of 40 patients per year over a 24 months enrolment period. Criteria for defining sample size do not follow statistical power estimates in order to demonstrate difference between the alternative donor options.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Primary induction Failure or chemoresistant relapse in Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) patients

Activation of an alternative donor search by the Italian Bone Marrow Donor Registry (IBMDR)

Age >=18<=70

Unavailability of a HLA-matched related donor (MRD)

Performance status: ECOG<=3

Written and signed informed consent

Life expectancy not severely limited by concomitant illness.

Exclusion Criteria:

Previous allogeneic transplant (autologous transplant is accepted)

Positive pregnancy test

Any active, uncontrolled infection.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2 years from time of enrolment
  The overall survival at 2 years (from time of enrolment) of all patients enrolled in to the study (either transplanted or not).
  This is the simplest outcome, defined as the probability of survival irrespective of disease state at any point in time. Patients alive at their last follow-up are censored. It is analyzed by the Kaplan-Meier method, Log-Rank Test and parametric or semiparametric survival models.
Disease-Free Survival (DFS) | 2 years from enrolment
  DFS is defined as the probability of being alive free of disease at any point in time. Thus, death or disease relapse are treated as events (1). Patients alive and free of disease at their last follow-up are censored. The statistical methods for the analysis of DFS are the same as for OS (Kaplan-Meier curve, Log-Rank Test and survival models).
Relapse Incidence (RI) | 2 years from enrolment
  RI is defined as the probability of having had a relapse before time t. Death without experiencing a relapse is a competing event. The correct method of analysis is therefore the estimation of the Cumulative Incidence curve, comparable by the Gray Test and, for the multivariate analysis, the application of the proportional hazard model for the sub-distribution of competing risks, by Fine and Gray. In studying relapse, sometimes the interest is not only in the estimation of the cumulative incidence curve, but also in the estimation of the hazard ratios for comparing groups of patients. It is therefore common to apply also a survival (Cox or parametric) model considering relapse as an event and death without relapse as a censoring (the response time is given by the minimum between time to relapse and time to death without relapse; as usual, a patient who is alive and free of relapse is also censored).
Non-Relapse Mortality (NRM) | 2 years from enrolment
  It is defined as the probability of dying without previous occurrence of a relapse, which is a competing event. The same indications as for the analysis of RI apply.
Progression-Free Survival (PFS) | 2 years from enrolment
  It is defined as the probability of being alive with no indication of disease progression (relapse is considered as progression for patients in CR). It is analyzed by KaplanMeier curve, Log-Rank Test and parametric or non-parametric survival models.

SECONDARY OUTCOMES:
Haematopoietic Recovery | participants will be followed for the duration of hospital stay, an expected average of 30 days
  The day of engraftment is defined as the first day of 3 consecutive days with a persistent blood cell count above a predefined level:
  WBC 1 x 109/l PMN 0.5 x 109/l Platelets 50 x109 /l or 20x 10 9 /l Death without recovery is a competing event, while no engraftment at the last followup is to be considered as a censored observation. Relapse or disease progression could be considered (depending on the disease being studied) as further competing events: this must be discussed with the responsible physician.
Acute Graft-versus-Host Disease (aGvHD) | from date of transplant to until the date of first event of aCGVD assessed up to 100 days post transplant
  The available information in the EBMT data regard the date of onset and the maximum grade of aGvHD. It is therefore possible to estimate the probability of aGvHD in a competing risks setting (death is a competing event; whether relapse/progression is a competing event must be discussed with the physician). By definition, patients alive (relapse/progression-free) at day 100 without having experienced aGvHD are censored. If the dates of onset are missing for the majority of patients, the analysis can focus only on the occurrence of aGvHD, which is analyzed by a logistic regression model. This method would however be incorrect if there is a (non negligible) percentage of censored observations or if competing events occurred before day 100.
Chronic Graft-versus-Host Disease (cGvHD) | from day +100 post transplant to until the date of first event to cGVHD assessed up to 2 years post enrolment
  When possible, if information on the date of 1°occurrence of cGvHD is available, it should be analyzed as a time-to-event outcome, being death (and possibly relapse/progression) the competing event; data are censored for patients alive (relapse/progression-free) without episodes of cGvHD at last follow-up. Since cGvHD is defined only for patients surviving at least 100 days, the survival model should consider a left truncation at 100 days; alternatively, the time of occurrence of cGvHD must be computed from 100 days. If information on the timing of cGvHD is not available, the outcome considered is the occurrence, and the statistical model to be used is the logistic regression. Only patients surviving at least 100 days are considered to be at risk of developing cGvHD, therefore the analysis must be restricted to these patients. This analysis is of course not satisfactory because it does not take into account the occurrence of death and censoring.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — Ospedale San Raffaele
Locations (30):
- Italy (30):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Policlinico, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale San Orsola, Bologna
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - Ospedale Binaghi, Cagliari
  - Ospedale Oncologico Businco, Cagliari
  - Ospedale Ferrarotto - Ematologia, Catania
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ospedale Policlinico San Martino - IST, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Niguarda Ca' Grande, Milan
  - Ospedale San Raffaele, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - Cattedra di Medicina Interna ed Ematologia - Ospedale S. Gerardo de' i Tintori - Università degli Studi di Milano, Monza
  - AO Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Dipartimento Oncologico La Maddalena, Palermo
  - Fondazione IRCCS San Matteo, Pavia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Cattedra di Ematologia - Policlinico, Roma
  - Policlinico A. Gemelli, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - U.O. di Ematologia e Trapianti di Midollo Osseo - Azienda Osp. S. Camillo-Forlanini / Padiglione Morgagni, Roma
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale San Giuseppe Moscato, Taranto
  - Azienda ospedaliera Città della Salute e della Scienza, Torino
  - Centro Trapianti Metropolitano, Torino
  - A.O. Santa Maria della Misericordia, Udine